CLINICAL TRIAL: NCT01273805
Title: Phase II Study of Hydroxychloroquine in Previously Treated Patients With Metastatic Pancreatic Cancer
Brief Title: Hydroxychloroquine in Previously Treated Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Brian Wolpin, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-310
Record Dates: First submitted 2011-01-07; First posted 2011-01-11 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Pancreatic Cancer
Keywords: metastatic pancreatic cancer; hydroxychloroquine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: There were 2 arms in this study because the study was amended to evaluate a second cohort of patients treated at a higher dose using the same two-stage statistical design.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxychloroquine 400 mg b.i.d. (Experimental): Patients received 400 mg hydroxychloroquine orally twice per day. Cycle duration was 4 weeks. Patients remained on treatment indefinitely without the occurrence of disease progression, unacceptable adverse events, patient withdrawal, or discontinuation per MD decision.
  Interventions: Drug: Hydroxychloroquine
- Hydroxychloroquine 600 mg b.i.d. (Experimental): Patients received 600 mg hydroxychloroquine orally twice per day. Cycle duration was 4 weeks. Patients remained on treatment indefinitely without the occurrence of disease progression, unacceptable adverse events, patient withdrawal, or discontinuation per MD decision.
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine
  Other Names: Plaquenil

SUMMARY:
Hydroxychloroquine is approved for the treatment of non-cancerous illnesses such as rheumatoid arthritis and systemic lupus erythematous. Researchers in the laboratory have tested tumors from patients with pancreatic cancer and have discovered that they have certain pathways inside the cells that promote growth and survival of the tumor. Hydroxychloroquine may inactivate these pathways and results in the death of pancreatic cancer cells.

DETAILED DESCRIPTION:
Primary Objective

* To determine the efficacy of single-agent hydroxychloroquine in patients with metastatic pancreatic cancer previously treated with one or two prior chemotherapy regimens as measured by progression-free survival at two months

Secondary Objectives

* To assess tumor response rate, biochemical response rate (i.e. decrease in serum CA19-9 by > 30%), and overall survival

Translational/Exploratory Objectives

* To investigate predictors of response to anti-autophagy therapy with hydroxychloroquine
* To explore the kinetics of in vivo autophagy inhibition using peripheral blood WBCs to monitor autophagic activity among patients receiving hydroxychloroquine

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable pancreatic adenocarcinoma that is metastatic to distant sites
* Measurable disease, defined as at least one lesion that can accurately be measured in at least one dimension
* Patients must have been treated with one or two previous lines of chemotherapy for metastatic disease with documented tumor progression or intolerance due to toxicity
* Minimum of two weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy
* 18 years of age or older
* Life expectancy of greater than 12 weeks
* ECOG performance status of 0, 1 or 2
* Normal organ and marrow function as outlined in the protocol
* Patients must be able to swallow pills
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* More than two previous chemotherapy regimens for the treatment of metastatic pancreatic cancer
* Uncontrolled brain or leptomeningeal metastases
* History of macular degeneration, visual field changes, retinal disease, or cataracts that would interfere with funduscopic eye examinations
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to hydroxychloroquine
* Previous treatment with chloroquine or hydroxychloroquine for other indications, such as rheumatoid arthritis, SLE or malaria prophylaxis
* Prior treatment with any investigational drug within the preceding 4 weeks
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter absorption of hydroxychloroquine. Patients who have undergone a Whipple procedure for localized pancreatic cancer are not excluded from enrollment
* History of non-compliance to medical regimens
* Known diagnosis of glucose-6-phosphate deficiency, porphyria or psoriasis
* Penicillamine use for Wilson's disease or any other indication
* Uncontrolled intercurrent illness including but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3-years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past three years: cervical cancer in situ, and basal cell or squamous cell carcinoma
* HIV-positive individuals on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Wolpin, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wolpin BM, Rubinson DA, Wang X, Chan JA, Cleary JM, Enzinger PC, Fuchs CS, McCleary NJ, Meyerhardt JA, Ng K, Schrag D, Sikora AL, Spicer BA, Killion L, Mamon H, Kimmelman AC. Phase II and pharmacodynamic study of autophagy inhibition using hydroxychloroquine in patients with metastatic pancreatic adenocarcinoma. Oncologist. 2014 Jun;19(6):637-8. doi: 10.1634/theoncologist.2014-0086. Epub 2014 May 12. PMID 24821822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 participants were enrolled between January 2011 and October 2012.
Period: Overall Study
Arm/Group | Hydroxychloroquine 400 mg b.i.d. | Hydroxychloroquine 600 mg b.i.d.
Started | 10 | 10
Completed | 0 | 0
Not Completed | 10 | 10
Not completed — Radiologic PD or Symptom Deterioration | 10 | 10

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine 400 mg b.i.d. | Hydroxychloroquine 600 mg b.i.d. | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Full Range); unit: years] | 67.5 [56 to 83] | 66 [58 to 76] | 67 [56 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
ECOG Performance Status (PS) [Number; unit: participants] — ECOG PS0: Fully active, able to carry on all pre-disease performance without restriction ECOG PS1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG PS2: Ambulatory and capable of all self-care but unable to carry out any work activities; Up and about more than 50% of waking hours
  participants
    PS0 | 1 | 1 | 2
    PS1 | 5 | 8 | 13
    PS2 | 4 | 1 | 5
Site of Primary Tumor [Number; unit: participants]
  Head or Head and Body | 6 | 7 | 13
  Body or Tail | 4 | 3 | 7
Location of Metastasis [Number; unit: participants]
  Liver | 8 | 7 | 15
  Lung | 4 | 3 | 7
  Peritoneum | 4 | 5 | 9
  Other | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: 2-month Progression-Free Survival Rate
Description: 2-month progression-free survival rate was defined as the percentage of patients absent progression (PD) or death before 2 months. Patients were considered to have experienced PD if they demonstrated either clinical deterioration resulting in withdrawal or PD per RECIST 1.0 criteria: At least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and at the first restaging at 2 months.
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Hydroxychloroquine 400 mg b.i.d. | Hydroxychloroquine 600 mg b.i.d.
Number analyzed (Participants) | 10 | 10
percentage of patients | 10 [.28 to 44.5] | 10 [.28 to 44.5]

2. Secondary Outcome: Biochemical Response Rate
Description: Biochemical response rate was defined as the percentage of patients achieving on treatment a decrease in serum CA 19-9 by > 30% from baseline.
Time Frame: Disease was evaluated radiologically at baseline and every 2 months on treatment. Median duration of treatment for this study cohort was 34 days.
Population: Biochemical response could not be estimated due to insufficient longitudinal CA 19-9 measurements. This was directly related to the observed lack of activity of the study drug and corresponding short duration of therapy.
Arm/Group | Hydroxychloroquine 400 mg b.i.d. | Hydroxychloroquine 600 mg b.i.d.
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Tumor Response Rate
Description: Tumor response rate is the percentage of patients achieving complete or partial response on treatment based on RECIST 1.0 criteria. For target lesions, complete response (CR) is disappearance of all target lesions and partial response (PR) is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. CR for the evaluation of non-target lesions is the disappearance of non-target lesions and normalization of tumor marker level. Appearance of one or more new lesions is classified as progression of non-target lesions. CR or PR confirmation is required >/= 4 weeks.
Time Frame: as for outcome 2
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Number; unit: percentage of patients
Arm/Group | Hydroxychloroquine 400 mg b.i.d. | Hydroxychloroquine 600 mg b.i.d.
Number analyzed (Participants) | 10 | 10
percentage of patients | 0 | 0

4. Secondary Outcome: Overall Survival
Description: Overall survival estimated using Kaplan-Meier (KM) methods is defined as the time from study entry to death or date last known alive.
Time Frame: All patients were followed until death. Median survival follow-up in this study cohort was 60 days (95% CI: 40-184).
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Hydroxychloroquine 400 mg b.i.d. | Hydroxychloroquine 600 mg b.i.d.
Number analyzed (Participants) | 10 | 10
days | 51.5 [24 to 275] | 83 [40 to 178]

5. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to time of objective progression on CT scan or the time of death for patients with clinical deterioration resulting in withdrawal from the trial. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions. Patients without an event were censored at date of last disease evaluation.
Time Frame: Disease was evaluated radiologically at baseline and every 2 months on treatment. Median PFS follow-up in this study cohort was 46.5 days (95% CI 33-61).
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Hydroxychloroquine 400 mg b.i.d. | Hydroxychloroquine 600 mg b.i.d.
Number analyzed (Participants) | 10 | 10
days | 51.5 [16 to 66] | 44.5 [33 to 74]

6. Secondary Outcome: Grade 4-5 Treatment-Related Toxicity
Description: All grade 4-5 adverse events with treatment attribution of possibly, probably or definite based on CTCAEv3 as reported on case report forms.
Time Frame: Adverse events were assessed each cycle throughout treatment. Participants were followed for the duration of treatment, an average of 34 days for this study population.
Population: The analysis dataset is comprised of all treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine 400 mg b.i.d. | Hydroxychloroquine 600 mg b.i.d.
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were assessed each cycle throughout treatment. Participants were followed for the duration of treatment, an average of 34 days for this study population.
Description: Maximum grade toxicity by type for a patient over time including only treatment-related events (possible, probable or definite attribution) was first calculated with patients therefore appearing once for a given type of toxicity. Serious and Other AEs were defined as events of grades 3-5 and grades 1-2, respectively, based on CTCAEv3.
Arm/Group | Hydroxychloroquine 400 mg b.i.d. | Hydroxychloroquine 600 mg b.i.d.
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydroxychloroquine 400 mg b.i.d. (N=10) | Hydroxychloroquine 600 mg b.i.d. (N=10)
Elevated alanine aminotransferase (Investigations) | 1 | 0
lymphopenia (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydroxychloroquine 400 mg b.i.d. (N=10) | Hydroxychloroquine 600 mg b.i.d. (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 2
Blurred vision (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 5
Elevated alanine aminotransferase (Investigations) | 1 | 0
Elevated alkaline phosphatase (Investigations) | 3 | 0
Elevated aspartate aminotransferase (Investigations) | 3 | 0
Facial edema (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Hyperbilirubinemia (Investigations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Leukopenia (Investigations) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash, maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No